CLINICAL TRIAL: NCT06182891
Title: Department of Pharmacy, the Affiliated Hospital of Xuzhou Medical University
Brief Title: Renoprotective Effects of Dulaglutide in Patients With Type 2 Diabetic Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2021-KL236-02
Record Dates: First submitted 2023-11-07; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetic Nephropathy
Keywords: dulaglutide; diabetic nephropathy; renoprotective effects
MeSH Terms: conditions — Diabetic Nephropathies | interventions — dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dulaglutide (Experimental): Dulaglutide was injected subcutaneously at standard dose and frequency for consecutive 12 months.
  Interventions: Drug: Dulaglutide Injection
- other hypoglycemic agents not including GLP-1 receptor agonists (Active Comparator): Other hypoglycemic agents not including GLP-1 receptor agonists were used at standard dose and frequency for consecutive 12 months.
  Interventions: Drug: Dulaglutide Injection

INTERVENTIONS:
Drug: Dulaglutide Injection — Dulaglutide injection was injected subcutaneously at standard dose and frequency for consecutive 12 months in patients with type 2 diabetes and diabetic kidney disease. Other hypoglycemic agents not including GLP-1 receptor agonists were used at standard dose and frequency for consecutive 12 months.
  Other Names: Other hypoglycemic agents not including GLP-1 receptor agonists

SUMMARY:
The purpose of the real-world observational prospective study is to access the renoprotective effects of dulaglutide as well as to explore corresponding mechanisms in patients with Type 2 Diabetic Nephropathy.

DETAILED DESCRIPTION:
Related studies have found that Glucagon-like peptide-1 (GLP-1) receptors are localized on a variety of tissues and cell types in addition to pancreatic β-cells, and GLP-1 and GLP-1 receptor agonists can exert diverse effect on multiple organs and tissues, with pleiotropic potential physiological, pathophysiological as well as pharmacological implications. Multiple clinical trials suggest that GLP-1 receptor agonists can exert renoprotective effects and persuasively inhibit the progression of kidney disease in type 2 diabetic patients. The beneficial effects of GLP-1 receptor agonists on Type 2 Diabetic Nephropathy, independent of their hypoglycemic ability, might are mediated by anti-oxidative stress, anti-inflammatory and natriuresis properties. However, it is not clear whether the above-mentioned properties are involved in the EMT process of renal tubular epithelial cells.

All participants meeting all eligibility criteria received routine medical consultations. During routine medical visits, patients were randomized into two groups (1.07:1) to receive a total duration of 12 months of hypoglycemic therapy - dulaglutide plus other hypoglycemic agents not including GLP-1 receptor agonists (intervention group), and other hypoglycemic agents not including GLP-1 receptor agonists (control group). A random number method was applied for grouping in this study. Dulaglutide and other hypoglycemic agents were administered according to the drug package insert. Of course, the investigators decided on other background treatments for hypertension, hyperlipidemia, or cardiovascular-related risk factors based on the latest guidelines throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* All adults aged 18 and above
* No minors involved in the study
* Diabetic Nephropathy defined as a urinary albumin-to-creatinine ratio ≥30 mg/g at least twice in three measurements within a period of 3-6 months

Exclusion Criteria:

* Patients with other types of kidney disease
* Urinary tract infection
* Type 1 diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the urinary albumin-to-creatinine ratio | 3,6 and 12 months after dulaglutide injection treatment
  the changes in the urinary albumin-to-creatinine ratio
Evaluation of the biomarkers of the epithelial-mesenchymal transition process | 3,6 and 12 months after dulaglutide injection treatment
  the changes in the biomarkers of the epithelial-mesenchymal transition process from the baseline at 3, 6 and 12 months. These biomarkers of the epithelial-mesenchymal transition process include E-cadherin and periostin.

SECONDARY OUTCOMES:
Evaluation of the estimated glomerular filtration rate | 3,6 and 12 months after dulaglutide injection treatment
  the changes in the estimated glomerular filtration rate
Evaluation of the cystatin C | 3,6 and 12 months after dulaglutide injection treatment
  the changes in the cystatin C
Evaluation of adverse event | 3,6 and 12 months after dulaglutide injection treatment
  Tolerability and safety outcomes included the incidence of hypoglycemia, gastrointestinal reaction and other adverse events, which were recorded in detail at follow-up (3,6 and 12 months after dulaglutide injection treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Renhao Wang, Ph.D, Study Director — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- Department of Endocrinology, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952